CLINICAL TRIAL: NCT04717830
Title: An Open Study of the Safety and Pharmacokinetics of a Drug for the Emergency Prevention of Ebola Virus Disease Based on Humanized Monoclonal Antibodies
Brief Title: An Open Study of the Safety and Pharmacokinetics of a Drug for the Emergency Prevention of Ebola Virus Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-AT-2020
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gamezumab 1/10 therapeutic dose (Experimental): 1/10 therapeutic dose (5 volunteers)
  Interventions: Drug: Gamezumab
- Gamezumab 1/2 therapeutic dose (Experimental): 1/2 therapeutic dose (5 volunteers)
  Interventions: Drug: Gamezumab
- Gamezumab full therapeutic dose (Experimental): therapeutic dose (10 volunteers)
  Interventions: Drug: Gamezumab

INTERVENTIONS:
Drug: Gamezumab — solution for infusion
  Other Names: monoclonal antibodies against Ebola virus disease

SUMMARY:
Open-label safety, tolerability, pharmacokinetics and immunogenicity study in three dose escalation groups

DETAILED DESCRIPTION:
This Phase I clinical trial was developed to study drug safety, tolerability, and pharmacokinetics of the medicine for Ebola fever emergency prevention based on monoclonal recombinant antibodies in single use in healthy volunteers with a dose escalation. A consecutive recruitment of people who signed the Informed Consent Form into three groups of volunteers with different drug doses is made according to the volunteers' screening results. The total number of volunteers receiving the drug will be not less then 25 people.The purpose of this study is to assess safety, tolerability, and pharmacokinetics of a medicine for Ebola fever emergency prevention based on monoclonal recombinant antibodies in a single dose in healthy volunteers.

The study will include volunteers of both sexes, aged 18 to 45 years inclusive. Only 25 people will take part in the study and will receive the study drug, of which 5 will receive 1/10 of the therapeutic dose, 5 - 1/2 of the therapeutic dose, 15 - in the full therapeutic dose.

Participation of 5 doubles is envisaged: 1 person for a group of 5 volunteers and 3 for 15.

ELIGIBILITY:
Inclusion Criteria:

-• Availability of written Informed Consent to participate in the research;

* Men and women between the ages of 18 and 45;
* Absence in the history, as well as according to the screening examination of pathology from the gastrointestinal tract, liver, kidneys, cardiovascular system, central nervous system, musculoskeletal system, genitourinary, immune and endocrine systems, blood, which can affect the safety of the volunteer and the assessment of the research results (clinical, instrumental and laboratory studies did not reveal diseases or clinically significant abnormalities);
* Consent to use effective contraceptive methods during the entire period of participation in the study
* Body mass index (BMI) is 18.5≤ BMI≤30;
* Absence of acute infectious diseases at the time of drug administration and 14 days before drug administration;
* Absence of allergic diseases in anamnesis
* No history of pronounced complications from previous use of immunobiological drugs;
* Negative pregnancy test based on urine test results (for women of childbearing age);
* Negative tests for HIV, hepatitis B and C, syphilis;
* Negative test for the presence of drugs and psychostimulants in the urine;
* Negative test for alcohol content;
* Indicators of general and biochemical analysis of blood, immunoglobulin E at screening within 1.1 X upper limit of the reference interval- 0.9 X lower limit of the reference interval
* Absence of changes in the myocardium of an inflammatory or dystrophic nature according to the results of ECG at screening

Exclusion Criteria:

* Participation of a volunteer in any other research within the last 90 days;
* Acute infectious and non-infectious diseases, exacerbations of chronic diseases during the 4 weeks preceding the screening;
* Vaccination against Ebola virus disease with any drugs, or administration of monoclonal antibodies against Ebola virus disease, including in the course of other clinical trials
* Treatment with steroids (except for hormonal contraceptives) in the last 10 days;
* Administration of immunoglobulins or other blood products in the last 3 months;
* Taking immunosuppressive drugs and / or immunomodulators within 6 months before the start of the study;
* Pregnancy or breastfeeding;
* Systolic blood pressure less than 100 mm Hg. or above 139 mm Hg; diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg; heart rate less than 60 beats / min or more than 100 beats / min;
* Aggravated allergic anamnesis (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, atopy, a history of serum sickness, hypersensitivity or allergic reactions to the administration of immunobiological drugs, known allergic reactions to the drug components, etc.), IgE total at the screening visit more than 2x upper limit of the reference interval;
* Diabetes mellitus or other forms of impaired glucose tolerance;
* The presence of a concomitant disease that may affect the assessment of the study results or which, in the opinion of the researcher, will not allow the volunteer to participate in the study or may affect the study and / or its results (including the assessment of safety parameters);
* A history of malignant neoplasms;
* Donation of blood (450 ml or more of blood or plasma) less than 2 months before the start of the study;
* Taking narcotic and psychostimulating drugs at the present time or in history;
* Alcohol intake in excess of the low risk level: no more than 20 grams of pure alcohol per day, no more than 5 days a week, alcohol intake within 48 hours before the administration of the study drug;
* Smoking: more than 10 cigarettes a day;
* Planned hospitalization and / or surgical intervention during the period of participation in the study, as well as 4 weeks before the expected date of drug administration.
* The presence of a concomitant disease that may affect the assessment of research results
* The volunteer's weight is less than 45 and more than 100 kg (even if the BMI of the volunteer meets the norm - clause 5 of the inclusion criteria)
* Any condition that, in the opinion of the investigator's physician, may be a contraindication to participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Serious Adverse Events | through the whole study, an average of 90 days
  Determination of Number of Participants With Serious Adverse Events
Number of Participants with Solicited Local and Systemic Adverse Events | through the whole study, an average of 90 days
  Determination of Number of Participants with Solicited Local and Systemic Adverse Events
Pharmacokinetics Study | before drug administration, after 1, 4, 8, 24, 36 and 48 hours after drug administration, and 7, 10, 14, 21, 28, 45, 60 and 90 days study.
  Immunological methods will be used to study the level of specific antibodies (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Zubkova, Principal Investigator — Research Institute of Influenza, Sankt-Peterburg, Russian Federation
Locations (1):
- Research Institute of Influenza, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No